CLINICAL TRIAL: NCT03095742
Title: Bedside Monitoring of Cerebral Energy State During the Peri-cardiac Arrest Period - Blood Pressure Targets in Post Resuscitation Care
Brief Title: Bedside Monitoring of Cerebral Energy State During the Peri-cardiac Arrest Period
Acronym: MICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Simon Mölström, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: S-20150173 HLP
Record Dates: First submitted 2017-03-17; First posted 2017-03-30 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Cardiac Arrest; Neurological Complication; Post-Cardiorespiratory Arrest Coma
Keywords: Microdialysis; Cerebral metabolism; Cardiac arrest; Intravenous; Neurological prognosis
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Single center randomized trial with allocation of 60 comatose out-of-hospital cardiac arrest patients undergoing TTM, to normal or high blood pressure target during ICU stay. Secondary a descriptive prospective cohorte study, measuring LP ratio obtained by microdialysis (MD) of the cerebral venous outflow, during the peri-cardiac arrest period
Who Masked: Participant, Care Provider, Investigator
Masking Description: Interventions are considered emergency procedures and study blood pressure measurement using the study blood pressure modules should be commenced as soon as possible after sustained ROSC, screening and randomisation. Study target blood pressure will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low MAP (Placebo Comparator): Low mean arterial pressure. 30 patients were blindly randomized to normal range (MAP 65 mmHg) during the peri-cardiac arrest period.
  Interventions: Diagnostic Test: Low MAP
- High MAP (Active Comparator): High mean arterial pressure. 30 patients were blindly randomized to intervention group (MAP 75 mmHg) during the peri-cardiac arrest period.
  Interventions: Diagnostic Test: High MAP

INTERVENTIONS:
Diagnostic Test: Low MAP — Extracerebral MD catheters were positioned in a retrograde direction in the internal jugular vein
  Other Names: Intravenous microdialysis
  Arms: Low MAP
Diagnostic Test: High MAP — Extracerebral MD catheters were positioned in a retrograde direction in the internal jugular vein
  Other Names: Intravenous microdialysis
  Arms: High MAP

SUMMARY:
In comatose patients resuscitated from out of hospital cardiac arrest (OHCA), neurological injuries remain the leading cause of death. The in-hospital mortality is reported at 30-50%, and the total mortality, although improved substantially over the last decade, remain to be significant, in most countries at up to 90%. An adequate blood pressure must be maintained in the post-cardiac arrest patient and helps to avoid further brain injury. The current trial addresses strategies for neuroprotection using a design of two different target blood pressure levels. "Normal MAP" (approximately 65 mmHg) vs. "high MAP" (approximately 75 mmHg). Markers measuring global cerebral ischemia caused by cardiac arrest and consecutive resuscitation, and reflecting the metabolic changes after successful resuscitation are urgently needed to enable a more personalized resuscitation and post resuscitation care.

It is technically simple and feasible to place a microdialysis catheter in the jugular bulb and monitor biochemical variables related to cerebral energy metabolism bedside. The LP ratio obtained from microdialysis of cerebral venous blood may be a sensitive indicator of impending cerebral damage and might play a critical role in detecting the early responses of post resuscitation care. Aim of this study is to investigate the global cerebral metabolic changes during CA and post-resuscitation care.

DETAILED DESCRIPTION:
Microdialysis assessment of cerebral energy state during cardiac arrest and cardiopulmonary resuscitation in humans

In comatose patients resuscitated from out of hospital cardiac arrest (OHCA), neurological injuries remain the leading cause of death. The in-hospital mortality is reported at 30-50%, and the total mortality, although improved substantially over the last decade, remain to be significant, in most countries at up to 90%. The brain of a patient resuscitated after cardiac arrest (CA) may have suffered ischemia and when spontaneous circulation is re-established, the subsequent reperfusion may cause further damage. Brain ischemia and the reperfusion injury lead to tissue degeneration and loss of neurological function, the extent dependent on duration and density of the insult. Temperature control and Targeted Temperature Management (TTM) targeting 33-36°C may mitigate this damage and is recommended in current international guidelines. However, managing post cardiac arrest patients are much more complicated than TTM alone, and blood pressure measurements and mechanical ventilation as part of post resuscitation care is emphasized. An adequate blood pressure must be maintained in the post-cardiac arrest patient. Episodes of hypotension can cause secondary injury, in addition to any initial insult incurred during the arrest by the brain and other organs. Mean arterial blood pressure (MAP) should be above 65 mmHg to reverse the acute shock state, and may preferably 80 to 100 mmHg to optimize cerebral perfusion. When determining blood pressure goals, clinicians must balance the metabolic needs of an ischemic brain with the potential for overstressing a decompensated heart. Cerebral autoregulation is often impaired after cardiac arrest, and brain perfusion declines when the MAP falls below 80 to 100 mmHg. Thus, maintaining an adequate MAP helps to avoid further brain injury. However, blood pressure goals have not been investigated in prospective clinical trials, and remain to be based on observational data and extrapolation from experimental data. While experimental studies suggest that high mean blood pressure targets are needed for maintaining cerebral blood flow, registries on consecutive clinical cases undergoing post resuscitation care suggest that lower blood pressure targets are used in clinical practice. But data RCT´s addressing specific targets in post resuscitation care have not been performed. The current trial addresses these strategies for neuroprotection in using design of two different target blood pressure levels. Intervention: 1:1 randomization:

"Normal MAP" (approximately 65 mmHg) vs. "high MAP" (approximately 75 mmHg) Markers measuring global cerebral ischemia caused by cardiac arrest and consecutive resuscitation, and reflecting the metabolic changes after successful resuscitation are urgently needed to enable a more personalized resuscitation and post resuscitation care.

It is technically simple and feasible to place a microdialysis catheter in the jugular bulb and monitor biochemical variables related to cerebral energy metabolism bedside. The LP ratio obtained from microdialysis of cerebral venous blood may be a sensitive indicator of impending cerebral damage and might play a critical role in detecting the early responses of post resuscitation care. Aim of this study is to investigate the global cerebral metabolic changes during CA and post-resuscitation care.

Aim: The study aim to (I) investigate whether the LP ratio obtained by microdialysis (MD) of the cerebral venous outflow reflects a derangement of global cerebral energy state during the peri-cardiac arrest period and (II) investigate the correlation between LP ratio and neurological outcome among patients with cardiac arrest and (III) investigate the correlation between LP ratio and the randomized blood pressure targets.

Design: The trial was a sub-study in the Blood Pressure and Oxygenation Targets after Out-of-Hospital Cardiac Arrest-trial (BOX, clinicaltrials.gov NCT03141099). This single center randomized trial allocated 60 comatose out-of-hospital cardiac arrest patients undergoing TTM, to normal or high blood pressure target during ICU stay. Secondary a descriptive prospective cohorte study, measuring LP ratio obtained by microdialysis (MD) of the cerebral venous outflow, during the peri-cardiac arrest period.

Primary outcome: Analysis will compare the two target blood pressure groups with respect to LP ratio.

Secondary outcomes: Cerebral Performance Category (CPC) when discharged from hospital, time to death, daily cumulated vasopressor requirement during ICU stay and need for combination of vasopressors and inotropic agents or mechanical circulatory support. All end-points are correlated to the randomized blood pressure groups. A stratified analysis by the following pre-defined design variables will also be performed: sex, age above median, median time to ROSC, known hypertension, known COPD, shockable primary rhythm.

Method: Interventions are considered emergency procedures and study blood pressure measurement using the study blood pressure modules should be commenced as soon as possible after sustained ROSC, screening and randomisation. Study target blood pressure will be blinded. Patients will be mechanically ventilated, sedated (propofol/fentanyl) and when necessary paralysed with neuromuscular blocking agents to reduce shivering and subsequent heat-generation and energy consumption. The core body temperature will be set as quickly as possible at the predefined target temperature, according to intervention allocation, with 4°C intravenous solutions, and commercially available cooling devices at the discretion of the treating physician. The target core temperature is then maintained for 24 h. After the maintenance period core temperature is gradually raised to normothermia of 37°C with a rewarming rate of no more than 0.5°C/hour. Body temperature is then maintained at normothermia 37 ±0.5°C for as long the as patient is comatose until 72 hours from sustained ROSC in treatment groups, using pharmacological treatment and temperature management systems when applicable.

The study is targeting low-normal paO2 of 9.5 kPa during TTM and when mechanical ventilation is needed. The target PaO2 is reached by adjusting FiO2 and PEEP on the ventilator as long as the patient in on controlled ventilation. Patients ventilation is adjusted, targeting normocapnia of paCO2 of 4,5 - 6,0 in all patients. Serial arterial blood gas analyses will be performed open label using the commercially available equipment adjusted to 37 °C (alpha-stat).

MD catheter (CMA 67, MDialysis AB, Stockholm, Sweden) is placed in a retrograde direction into the jugular bulb. A second identical MD catheter is inserted into one brachial artery. Both catheters are inserted through a peripheral intravenous 17 GA cannula using ultrasound guidance. The positioning of the catheter in the jugular bulb above the inlet of the common facial vein is verified on lateral neck radiograph according to accepted principles. MD catheters are perfused by MD pumps (CMA 106, MDialysis AB, Stockholm, Sweden) at 0.3 μL/min. The perfusates are collected in microvials and analyzed every one hour for 72 hours by enzymatic photometric techniques and displayed bedside (Iscus, Mdialysis AB, Stockholm, Sweden). The analyses include the variables routinely monitored during intracerebral microdialysis: glucose, pyruvate, lactate, glutamate and glycerol.

Neurological status, according to the CPC-scale, and survival are evaluated every day in the intensive care unit and/or at day 1, 2, 3, 4, 5, 6, 7 and at hospital (including local hospital) discharge, whichever comes first.

The Danish Regional Committee on Health and Research Ethics approved the study. Trial registration: S-20150173 HLP.

Perspectives The prognosis of patients who are admitted in a comatose state following successful resuscitation after cardiac arrest remains uncertain. Although the introduction of therapeutic hypothermia (TH), targeted temperature management (TTM) and improvements in post-resuscitation care have significantly increased the number of patients who are discharged home with minimal brain damage, short-term assessment of neurological outcome remains a challenge. The need for early and accurate prognostic predictors is crucial, especially since sedation and TH/TTM may alter the neurological examination and delay the recovery of motor response for several days. The development of additional tools, including electrophysiological examinations (electroencephalography and somatosensory evoked potentials), neuroimaging and chemical biomarkers, may help to evaluate the extent of brain injury in these patients. Accurate prognostication of comatose patients treated with TH/TTM can be obtained only 72 to 96 hours after CA and requires a multimodal approach.

Markers measuring cerebral ischemia caused by cardiac arrest and consecutive resuscitation, and reflecting the metabolic changes after successful resuscitation are urgently needed to enable a more personalized resuscitation and post resuscitation care. The LP ratio obtained from microdialysis of cerebral venous blood may play a critical role in detecting the early responses of post resuscitation care, and may predict in hospital and long term prognosis in patients affected by brain injury after CA.

During the peri-cardiac arrest period the LP ratio obtained by microdialysis of the cerebral venous outflow may reflects a derangement of global cerebral energy state. The LP ratio obtained from microdialysis of cerebral venous blood in humans may be a sensitive indicator of impending cerebral damage among patients with cardiac arrest. Further, the study investigates the correlation between LP ratio and the randomized blood pressure targets. In the future this might optimize and individualize the management of post cardiac arrest patients.

Appendix:

Pre-defined methodological substudy conducted prior to the MICA-RCT:

This single-center prospective feasibility study explores the possibilities to use microdialysis (MD) for continuous monitoring of cerebral energy metabolism by analyzing the draining cerebral venous blood. Eighteen comatose patients (same inclusion criteria as MICA-study but without the MAP intervention) )will be continuously monitored with jugular bulb and radial artery (reference) MD following resuscitation. This feasibility study was designed to investigate whether bedside JBM reflects secondary brain injury after OHCA, and may be implemented as a clinical tool with implications for early prognosis and individualized treatment improving patient outcome. Therefore, we tested the hypothesis whether the lactate/pyruvate (LP) ratio monitored in the cerebral venous outflow reflected brain energy metabolism after cardiac arrest and hence was different from the LP ratio monitored in arterial blood.

The primary objective was to compare time-averaged means of microdialysis parameters (intervals of 12 hours) of the jugular venous and the arterial blood during post-resuscitation care. Secondary objectives of clinical interest were to compare (i) neuro-metabolic patterns between patients with unfavorable and favorable neurological outcome (ii) total duration of cerebral desaturation and clinical outcome.

Risks and discomforts: Few. The retrograde MD catheter is inserted under ultrasound guidance and is associated with a small (<2%) risk of localized bleed which can be managed by manual compression. Accidental arterial puncture occurs and is managed by manual compression. Strokes and air emboli are extremely rare and symptoms are usually transient. The blood drawn for blood gas analyses is not associated with increased risk, the volume needed is approximately 50 ml total and thus not associated with increased risks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Out-of-hospital cardiac arrest (OHCA)
* Presumed cardiac cause
* Unconsciousness (Glasgow Coma Score ≤8)
* Sustained return of spontaneous circulation (ROSC) (20 minutes of circulation)
* Target temperature management is indicated

Exclusion Criteria:

* Conscious patients
* Pregnancy
* OHCA of presumed non-cardiac cause
* Cardiac arrest after arrival in hospital
* Known bleeding diathesis
* Suspected or confirmed acute intracranial bleeding
* Suspected or confirmed acute stroke
* Temperature on admission <30°C
* Unwitnessed asystole
* Persistent cardiogenic shock
* Known limitations in therapy
* Known disease making 180 day survival unlikely
* Known pre-arrest cerebral performance category 3 or 4
* > 240 minutes from ROSC to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
LP ratio | Peri-caridac arrest period - 72 hours
  Analysis will compare the two target blood pressure groups with respect to lactate/pyruvate (LP) ratio.

SECONDARY OUTCOMES:
CPC | 72 hours
  Cerebral Performance Category (CPC) when discharged from hospital, time to death, daily cumulated vasopressor requirement during ICU stay and need for combination of vasopressors and inotropic agents or mechanical circulatory support..

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mølstrøm, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molstrom S, Nielsen TH, Nordstrom CH, Hassager C, Moller JE, Kjaergaard J, Moller S, Schmidt H, Toft P. Design paper of the "Blood pressure targets in post-resuscitation care and bedside monitoring of cerebral energy state: a randomized clinical trial". Trials. 2019 Jun 10;20(1):344. doi: 10.1186/s13063-019-3397-1. PMID 31182135